CLINICAL TRIAL: NCT00855010
Title: Effect of Pioglitazone on Pancreatic Steatosis and Bone Health
Brief Title: Pioglitazone on Pancreatic Steatosis and Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ildiko Lingvay, MD, MPH, MSCS, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112008-047; 1K23RRO24470-01; NCT00896116 (obsolete NCT alias)
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Pioglitazone; prediabetes; diabetes; obesity; Pancreatic fat
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pioglitazone (Experimental): pioglitazone tablet 45 mg once daily
  Interventions: Drug: pioglitazone
- placebo pill (Placebo Comparator): placebo pill once daily (look-alike pill which contains no active ingredients)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pioglitazone — pioglitazone 45 mg daily
  Other Names: Actos
  Arms: pioglitazone
Drug: placebo — one daily
  Other Names: Placebo tablet resembling pioglitazone 45 mg.
  Arms: placebo pill

SUMMARY:
Randomized, double blind, placebo controlled trial evaluating the effect of pioglitazone on pancreatic fat content and bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

* Fat level in the pancreas above 4% (measurement done by us with an MRI)
* English speaker
* over 21 years old

Exclusion Criteria:

* contraindication to MRI
* anemia
* pregnancy or desire to conceive
* use of unapproved medications
* prior pancreatic disease
* use of more then 2 alcoholic drinks every day

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone: pioglitazone tablet 45 mg once daily
  pioglitazone: pioglitazone 45 mg daily: 23 subjects
- Placebo Pill: placebo pill once daily (look-alike pill which contains no active ingredients)
  placebo: one daily: 19 subjects
Period: Overall Study
Arm/Group | Pioglitazone | Placebo Pill
Started | 23 | 19
Completed | 19 | 18
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone: pioglitazone tablet 45 mg once daily
  pioglitazone: pioglitazone 45 mg daily: 23
- Placebo Pill: placebo pill once daily (look-alike pill which contains no active ingredients)
  placebo: one daily: 19
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo Pill | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (9.9) | 52.2 (10.6) | 52.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 12 | 3 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Pancreatic Fat Content
Description: Pancreatic fat content was determined by proton magnetic resonance spectroscopy (1H-MRS) using a 1.5 Tesla Philips Intera system.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: Percentage of fat
Arm/Group | Pioglitazone | Placebo Pill
Number analyzed (Participants) | 23 | 19
Percentage of fat | 9.6 [5.1 to 16.6] | 13.0 [6.1 to 20.2]

2. Primary Outcome: Bone Turnover Marker - Intact Parathyroid Hormone (PTH)
Description: Intact parathyroid hormone (PTH) were measured using enzyme-linked immunosorbent assay. .
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Pioglitazone:: pioglitazone tablet 45 mg once daily
  pioglitazone: pioglitazone 45 mg daily
- Placebo Pill:: placebo pill once daily (look-alike pill which contains no active ingredients)
  placebo: one daily
Arm/Group | Pioglitazone: | Placebo Pill:
Number analyzed (Participants) | 23 | 19
pg/mL | 41 [38 to 57] | 56 [51 to 74]

3. Primary Outcome: Bone Turnover Marker - Plasma 25-hydroxyvitamin D
Description: Plasma 25-hydroxyvitamin D was determined by radioimmunoassay
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Pioglitazone | Placebo Pill
Number analyzed (Participants) | 23 | 19
ng/mL | 25 [15 to 30] | 19 [14 to 25]

4. Secondary Outcome: Beta-cell Function
Description: Changes in B-cell function as measured by acute insulin release to glucose (AIRg)
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: microUnits/mL x min
Arm/Group | Pioglitazone | Placebo Pill
Number analyzed (Participants) | 23 | 19
microUnits/mL x min | 101 [40 to 352] | 494 [264 to 748]

5. Secondary Outcome: Hepatic Fat Content
Description: Hepatic fat content was determined by proton magnetic resonance spectroscopy (1H-MRS) using a 1.5 Tesla Philips Intera system.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Pioglitazone | Placebo Pill
Number analyzed (Participants) | 23 | 19
percentage | 4.0 [1.7 to 10.9] | 5.8 [3.6 to 16.0]

6. Secondary Outcome: Subcutaneous Fat Area
Description: Abdominal MRI was performed to quantify subcutaneous fat area at the L2-L3 level.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Pioglitazone | Placebo Pill
Number analyzed (Participants) | 23 | 19
cm^2 | 243 (133) | 378 (179)

7. Secondary Outcome: Visceral Fat Area
Description: Abdominal MRI was performed to quantify visceral fat area at the L2-L3 level.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Pioglitazone | Placebo Pill
Number analyzed (Participants) | 23 | 19
cm^2 | 302 (88) | 273 (89)

8. Secondary Outcome: Bone Mineral Density
Description: Areal Bone Mineral Density at the L2-L4 antero-posterior lumbar spine, left femoral neck and total hip were measured by DXA scan using a Hologic Discovery Instrument scanner.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Pioglitazone | Placebo Pill
Number analyzed (Participants) | 23 | 19
g/cm^2
  L2-L4 Lumbar spine BMD | 1.03 (0.14) | 1.03 (0.14)
  Left femoral neck | 0.83 (0.09) | 0.85 (0.13)
  Left total hip | 0.96 (0.12) | 1.02 (0.12)

9. Secondary Outcome: Disposition Index
Description: Disposition index is a measure of insulin secretion multiplied by insulin sensitivity, both derived from intravenous glucose tolerance test. A higher number means the pancreas is better able to lower blood glucose and a lower number means the pancreas is less able to lower blood glucose
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: Unitless
Arm/Group | Pioglitazone: | Placebo Pill:
Number analyzed (Participants) | 23 | 19
Unitless | 410 [118 to 1458] | 841 [487 to 1491]

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Placebo Pill
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/19
Other Adverse Events (participants affected / at risk) | 7/23 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=23) | Placebo Pill (N=19)
Bacteremia with Streptococcus pneumoniae (Infections and infestations) | 1 (1) | 0 (0)
Motor vehicle trauma (Surgical and medical procedures) | 1 (1) | 0 (0)
Right ankle trauma (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=23) | Placebo Pill (N=19)
Lose consciousness (General disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fingers edema (General disorders) | 2 (2) | 1 (1)
Trauma (General disorders) | 2 (2) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Fatigue (Hepatobiliary disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lipoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No